CLINICAL TRIAL: NCT02225652
Title: A Phase II Study of Dose Density Regimen With Fluorouracil, Epirubicin and Cyclophosphamide at Days 1, 4 Every 14 Days With Filgrastim Support Followed by Weekly Paclitaxel in Women With Primary Breast Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST174.05; 2010-020772-38 (EudraCT Number)
Record Dates: First submitted 2014-08-25; First posted 2014-08-26 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Women With Primary Breast Cancer
MeSH Terms: interventions — FEC protocol; Fluorouracil; Epirubicin; Cyclophosphamide; Filgrastim; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FEC + filgrastim x 3 cycles q 14-21 days and Weekly Paclitaxel (Experimental): FEC (FLUOROURACIL 500 mg/m2 IV infusion of 30 minutes + EPIRUBICIN 60 mg/m2 IV infusion of 1 hour + CYCLOPHOSPHAMIDE 500 mg/m2 IV infusion of 30 minutes).
  From day 7 until hematological recovery = Filgrastim 300 microg s.c. After 21 days from the last FEC cycle = Paclitaxel 100 mg/m2 IV infusion of 1hour (weekly for 8 cycles, at day 1).
  Interventions: Drug: FEC (Fluorouracil, Epirubicin, Cyclophosphamide) + filgrastim + paclitaxel

INTERVENTIONS:
Drug: FEC (Fluorouracil, Epirubicin, Cyclophosphamide) + filgrastim + paclitaxel

SUMMARY:
TITLE: A Phase II Study of Dose Density Regimen with Fluorouracil, Epirubicin and Cyclophosphamide at Days 1, 4 Every 14 Days with Filgrastim Support followed by Weekly Paclitaxel in Women with Primary Breast Cancer.

PROTOCOL CODE: IRST 174.05

PHASE: II

STUDY DESIGN: Pharmacological, open-label, prospective, not randomized, monocentric trial

DESCRIPTION OF STUDY TREATMENT:

FEC + filgrastim x 3 cycles q 14-21 days

Day 1 and day 4 = FEC (FLUOROURACIL 500 mg/m2 IV infusion of 30 minutes + EPIRUBICIN 60 mg/m2 IV infusion of 1 hour + CYCLOPHOSPHAMIDE 500 mg/m2 IV infusion of 30 minutes).

From day 7 until hematological recovery = Filgrastim 300 microg s.c.

After 21 days from the last FEC cycle = Paclitaxel 100 mg/m2 IV infusion of 1hour (weekly for 8 cycles, at day 1).

NUMBER OF SUBJECTS: in the first stage, 11 patients have been planned, with an additional 27 patients to the second stage if at least 7 patients complete the planned treatment.

OBJECTIVES

Primary objective: this trial is designed to assess feasibility of the proposed regimen with regard to toxicity and deliverability. Tolerability is defined as absence of any grade 3 or higher nonhematologic toxicity (excluding alopecia, nausea/vomit, and bone pain, which might be a consequence of the administration of filgrastim). Deliverability is measured as the percentage of patients who complete the planned treatment.

Secondary objectives:

* Relapse-free survival: measured from enrollment to the first date between date of documented relapse (or death) or date of last tumor assessment (if no documented relapse), or the date of last tumor assessment before the start of any further antitumor therapy not planned in the protocol.
* Overall survival: measured from enrollment to the date of death of any cause or last follow-up.

CORRELATIVE/SPECIAL STUDIES: to evaluate retrospectively potential biomarkers of activity and toxicity of this regimen, blood and plasma samples until 15 mL each one will be collected at study entry, before first docetaxel administration and 3-4 weeks after last docetaxel administration. Moreover, a paraffin block or specimens of the primary tumor will be collected for biological studies.

STATISTICAL CONSIDERATIONS: This trial is designed to assess feasibility of the proposed regimen with regard to toxicity and deliverability.

Tolerability is defined as absence of any grade 3 or higher non-hematologic toxicity (excluding alopecia, nausea/vomit, and bone pain, which might be a consequence of the administration of filgrastim).

A Simon two-stage design has been used with a 60% tolerability rate considered not promising and an 80% tolerability rate as promising, and probability of type I and type II errors has been set to be 0.10.

In the first stage, 11 patients have been planned, with an additional 27 patients to the second stage if at least 7 patients complete the planned treatment. The regimen would be considered tolerable and worthy of further study if at the end of the trial 27 out 38 patients complete the planned treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed primary breast cancer
* Age ≥18 and < 70 years
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1 (see appendix B)
* >4 positive axillary nodes or high-risk breast cancer with <4 node-positive or node negative disease. Patients <4 node-positive or node negative disease are eligible if the tumor is >1cm and two or more of the following are present: histologic grade 3, Ki67>30%, estrogen receptor (ER) negativity, or lymphovascular invasion [39]
* Adequate hematological, hepatic and renal function, as follows: hemoglobin ≥ 9 g/dl, absolute neutrophil count ≥1,500/mL, platelets ≥100,000/mL, total bilirubin ≤1.5 x ULN, alkaline phosphatase, AST(SGOT) and ALT(SGPT) ≤ 2.5 x ULN (≤ 5 x ULN if liver metastases present), serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance >50 mL/min. Either INR or APTT < 1.5 x ULN;
* Known hormone receptor status (ER/PgR or ER alone);
* Must have received no other chemotherapy regimen.
* Baseline LVEF ≥55% measured by echocardiography
* No over expression and/or amplification of HER2 in the invasive component of the primary tumour (in case of neoadjuvant treatment, tissue sample used for HER2 testing should be collected before neoadjuvant treatment starts)
* Negative pregnancy test no more than 7 days before randomization; test pregnancy can be omitted only in women without any reproductive potential (e.g.: postmenopausal women, i.e. amenorrhoea ≥2 years or with previous hysterectomy or bilateral ovariectomy). Women of child-bearing potential must agree to use adequate contraception at the time of randomization and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician and coordinating centre (CC) immediately; women in lactation period must be excluded;
* Completion of all necessary baseline laboratory and radiological investigations
* Ability to understand and the willingness to sign a written informed consent document.
* Signed written informed consent

Exclusion Criteria:

* Metastatic disease
* Participation in another clinical trial with any investigational agents within 30 days prior to study screening.
* Contraindications or hypersensitivity to study drugs;
* Past (less than 10 years) or current history of malignant neoplasms, except for curatively treated 1) basal and squamous cell carcinoma of the skin or 2) carcinoma in situ of the cervix.

NOTE: Patients with a prior malignancy diagnosed greater than 10 years in the past who have been curatively treated with surgery ONLY, WITHOUT radiation therapy or systemic therapy (chemotherapy or endocrine) are eligible for the study. Patients with any prior diagnosis of invasive breast cancer or melanoma, at any time, are excluded from this study.

* Serious cardiac illness or medical conditions including but not confined to:

  * History of documented congestive heart failure (CHF) or systolic dysfunction (LVEF <55%);
  * High-risk uncontrolled arrhythmias (ventricular tachycardia, high-grade AV-block, supraventricular arrhythmias which are not adequately rate-controlled);
  * Angina pectoris requiring antianginal medication;
  * Clinically significant valvular heart disease;
  * Evidence of transmural infarction on ECG;
  * Poorly controlled hypertension (e.g. systolic >180mm Hg or diastolic >100mm Hg);
* Other concurrent serious diseases that may interfere with planned treatment including severe pulmonary conditions/illness;
* Any of the following abnormal laboratory tests immediately prior to randomisation:

  * serum total bilirubin >1.5 x upper limit of normal (ULN). In the case of known Gilbert's syndrome, a higher serum total bilirubin (<2 x ULN) is allowed
  * alanine amino transferase (ALAT) or aspartate amino transferase (ASAT) >2.5 x ULN;
  * alkaline phosphatase (ALP) >2.5 x ULN;
  * serum creatinine >2.0 x ULN;
  * total white blood cell count (WBC) <2.5 x 109/L;
  * absolute neutrophil count <1.5 x 109/L;
  * platelets <100 x 109/L.
* Malabsorption syndrome, any disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, or persons unable to swallow oral medication. Subjects with ulcerative colitis are also excluded;
* Pregnant, lactating or women of childbearing potential without a negative pregnancy test - urine or serum, within 7 days prior to randomization, irrespective of the method of contraception used, including tubal ligation.
* Women of childbearing potential, including women whose last menstrual period was <12 months ago (unless surgically sterile) who are unable or unwilling to use adequate contraceptive measures during study treatment. (adequate contraceptive measures are intra-uterine device, barrier method - condoms, diaphragm - also in conjunction with spermicidal jelly, or total abstinence. Oral, injectable or implant hormonal contraceptives are not allowed on this study)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-09; Primary Completion 2013-09 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Tolerability of the treatment | 18 months
  Tolerability is defined as absence of any grade 3 or higher non-hematologic toxicity (excluding alopecia, nausea/vomit, and bone pain, which might be a consequence of the administration of filgrastim).
Toxicity | 18 months
  All patients will be evaluated for toxicity according to NCI CTCAE v3.0 criteria. All patients will be evaluable for toxicity from the time of their first treatment. Safety analysis will be based on the population of all treated (at least one cycle) patients.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 18 months
  Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression.
Overall survival (OS) | 18 months
  Overall survival (OS) is defined as the duration of time from start of treatment to last follow-up visit or death.
Relapse-free survival | 18 months
  The relapse-free survival is measured from enrollment to the first date between date of documented relapse/progression (or death) or date of last tumor assessment (if no documented progression) or the date of last tumor assessment before the start of any further antitumor therapy not planned in the protocol.
Kaplan-Meier curves | 18 months
  Time related outcomes (PFS, OS) will be described using Kaplan-Meier curves. 95% Confidence Intervals for median time and for each year of follow-up will be calculated with non-parametric methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Irst, Meldola, FC, Italy

REFERENCES:
- [Derived] Pietri E, Andreis D, Fabbri F, Menna C, Schirone A, Kopf B, Rocca A, Amadori D, De Giorgi U. A phase II study of a dose-density regimen with fluorouracil, epirubicin, and cyclophosphamide on days 1 and 4 every 14 days with filgrastim support followed by weekly paclitaxel in women with primary breast cancer. Oncologist. 2015 Mar;20(3):239-40. doi: 10.1634/theoncologist.2014-0326. Epub 2015 Jan 30. PMID 25637379